CLINICAL TRIAL: NCT05990738
Title: DAREON™-9: A Phase Ib Open-label Dose Escalation and Dose Confirmation Safety Study of Intravenous BI 764532 in Combination With a Single Agent Chemotherapy for the Treatment of Patients With Relapsed/Refractory Small Cell Lung Cancer After Platinum-based Chemotherapy
Brief Title: DAREON™-9: A Study to Test How Well Different Doses of BI 764532 Are Tolerated by People With Small Cell Lung Cancer When Taken Together With a Single Agent Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0009; 2023-506007-26-00 (EU CTIS Number); U1111-1293-4098 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Carcinoma (SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: BI 764532 low dose + topotecan/single agent chemotherapy (Experimental)
  Interventions: Drug: BI 764532; Drug: Topotecan; Drug: Single agent chemotherapy
- Part A: BI 764532 medium dose + topotecan/single agent chemotherapy (Experimental)
  Interventions: Drug: BI 764532; Drug: Topotecan; Drug: Single agent chemotherapy
- Part A: BI 764532 high dose + topotecan/single agent chemotherapy (Experimental)
  Interventions: Drug: BI 764532; Drug: Topotecan; Drug: Single agent chemotherapy
- Part B: BI 764532 + topotecan (Experimental)
  Interventions: Drug: BI 764532; Drug: Topotecan

INTERVENTIONS:
Drug: BI 764532 — BI 764532
  Other Names: Obrixtamig
Drug: Topotecan — Topotecan
Drug: Single agent chemotherapy — single agent chemotherapy
  Arms: Part A: BI 764532 high dose + topotecan/single agent chemotherapy; Part A: BI 764532 low dose + topotecan/single agent chemotherapy; Part A: BI 764532 medium dose + topotecan/single agent chemotherapy

SUMMARY:
This study is open to adults with extensive stage small cell lung cancer. The study is in people with advanced cancer that had previously received platinum-based chemotherapy and are eligible to receive a single agent chemotherapy treatment.

The purpose of this study is to find the highest dose of BI 764532 that people can tolerate when taken together with a single agent chemotherapy. BI 764532 is an antibody-like molecule that may help the immune system fight cancer.

Participants may continue to take BI 764532 as long as they benefit from treatment and can tolerate it. During this time, participants visit the study site regularly. The visits also depend on the response to the treatment. At the study visits, the doctors check the health of the participants, take necessary laboratory tests, and note any health problems that could have been caused by the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years old and at least at the legal age of consent in countries where it is greater than 18 years at the time of signature of the informed consent form (ICF).
2. Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
3. Histologically or cytologically confirmed small cell lung cancer (SCLC). Patients with tumours with mixed histology are eligible only if SCLC component is predominant and represent at least 50% of the overall tumour tissue.
4. Extensive stage - small cell lung cancer (ES-SCLC) that progressed or recurred following platinum-based treatment, and anti- programmed cell death protein 1 (PD-1) or programmed cell death ligand 1 (PD-L1) as applicable.
5. Patients must be eligible for single agent chemotherapy treatment (used in the trial) according to label.
6. Availability of archival tumour tissue sample.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. Further inclusion criteria apply.

Exclusion Criteria:

1. Previous treatment in this trial.
2. Current enrolment in another investigational device or drug trial, or <30 days since ending another investigational device or drug trial(s).
3. Untreated or symptomatic brain metastases. Participants with treated, stable brain metastases are eligible provided they meet the following criteria:

   * Radiotherapy or major surgery for brain metastases was completed at least 2 weeks (for radiotherapy) or 4 weeks (for major brain metastases surgery) prior to the first administration of BI 764532.
   * Patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off anti-epileptic drugs for at least 7 days or on stable doses of anti-epileptic drugs for malignant central nervous system (CNS) disease.
4. Presence of leptomeningeal carcinomatosis.
5. Prior participation in clinical trials of BI 764532, including receiving standard of care in these trials OR prior treatment with T cell engager (TcE) or cell therapies targeting delta-like ligand 3 (DLL3).
6. Persistent toxicity from previous treatments that has not resolved to ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 (except for alopecia, asthenia/fatigue, CTCAE Grade 2 neuropathy, or Grade 2 endocrinopathies controlled by replacement therapy).
7. Major surgery (major according to the investigator's assessment) within 28 days prior to first administration of BI 764532 or planned during treatment period, e.g. hip replacement.
8. Previous or concomitant malignancies other than the one treated in this trial within the last 2 years except

   1. effectively treated non-melanoma skin cancers
   2. effectively treated carcinoma in situ of the cervix
   3. effectively treated ductal carcinoma in situ
   4. other effectively treated malignancy that is considered cured by local treatment Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Occurrence of dose limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | up to 9 weeks
Part B: Occurrence of DLTs during the on-treatment period | up to 36 months
Part B: Occurrence of AEs during the on-treatment period | up to 36 months

SECONDARY OUTCOMES:
Part A: Occurrence of DLTs during the on-treatment period | up to 36 months
Part A: Occurrence of AEs during the on-treatment period | up to 36 months
Part B: Objective response | up to 36 months
Part B: Duration of response | up to 36 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (6):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic - Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - East Carolina University, Greenville, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia
- France (3):
  - INS Curie, Paris
  - HOP Civil, Strasbourg
  - INS Gustave Roussy, Villejuif
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Polish Mother's Memorial Hospital - Research Institute, Lodz, Poland
- Leicester Royal Infirmary, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com